CLINICAL TRIAL: NCT02305199
Title: Comparison of Hartmann's Solution and Normal Saline on Postoperative Blood Glucose and Insulin Levels in Type II Diabetic Patients
Brief Title: Hartmann's Solution and Normal Saline in Type II Diabetes Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: impossible to enroll participants
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Associate Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YeungnamU
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Hartmann's solution
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hartmanns' solution (Active Comparator): All the participants went on a fast at midnight and 1 L of 5% dextrose fluid containing 10 units of regular insulin (RI) and 40 mEq of potassium was administered intravenously.
  On participant's arrival to the operation room, fluid from the ward was immediately removed and replaced it with 1 L of unknown fluid completely sealed in black bag. Neither the participant nor the researcher were aware of the type of the fluid.
  After the fluid change, general anesthesia was induced. Intraoperative blood glucose was checked every one hours and 20% dextrose was injected if the number was below 100 and RI was injected if the number was checked over 200.
  Interventions: Drug: Hartmann's solution
- Normal saline (Active Comparator): All the participants went on a fast at midnight and 1 L of 5% dextrose fluid containing 10 units of RI and 40 mEq of potassium was administered intravenously.
  On participant's arrival to the operation room, fluid from the ward was immediately removed and replaced it with 1 L of unknown fluid completely sealed in black bag. Neither the participant nor the researcher were aware of the type of the fluid.
  After the fluid change, general anesthesia was induced. Intraoperative blood glucose was checked every one hours and 20% dextrose was injected if the number was below 100 and RI was injected if the number was checked over 200
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hartmann's solution — Hartmann's solution containing 200 mg/L of calcium chloride, 300 mg/L of potassium chloride, 6 g/L of Sodium chloride, 3.1 g/L of Sodium lactate.
  Other Names: Hartmann solution 1000 ml, Choonwae pharmacy
  Arms: Hartmanns' solution
Drug: Normal saline — Fluid containing Sodium chloride 9 g/L
  Other Names: Normal Saline 1 L, Choonwae
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine whether perioperative use of Hartmann's solution in type II diabetes patients increases blood glucose level after surgery. The investigators expect the result to broaden the choice of fluid for diabetic patients and hopefully to diminish the side effects manifested by the excess use of normal saline.

DETAILED DESCRIPTION:
Hyperglycemia is an independent risk factor for poor outcomes in diabetic patients experiencing sudden cardiac death, myocardial infarction, cerebrovascular accident. During surgery, activation of the neuroendocrine system by surgical stress releases stress-induced hormones such as cortisol, glucagon, epinephrine, and growth hormones and it leads to hepatic glucogenesis and glycogenolysis. Acute perioperative hyperglycemia induces decreased microvascular reactivity to dilatory agents like bradykinin, increased inflammatory cytokines, and impaired neutrophil activity. This impaired neuroendocrine and immune system leads to increased inflammation and multiple organ system dysfunction.

Thomas and Alberti showed postoperative use of 1 litre of Hartmann's solution was associated with a 7.5 mmol/L increase in plasma glucose concentrations, compared with an increase of 2.1 mmol/L in diabetic patients who received no intravenous fluids. Since then, normal saline has been preferred over Hartmann's solution in fear of acute hyperglycemia during postoperative period.

However, a recent review suggested that the maximum increase in glucose concentration with 1 L of Hartmann's solution would be about 1 mmol/L (about 18 mg/dL) ,with a much lower effect on blood glucose in clinical practice.

In fact, according to 2012 National Health Services (NHS) diabetes guideline for the perioperative management of the adult patient with diabetes, Hartmann's solution is used in preference to 0.9% saline. Excess use of normal saline could yield complications such as hyperglycemia and metabolic acidosis.

To date, a few studies have examined the effects of preoperative blood glucose levels on outcomes in patients undergoing surgery, and no prospective randomized investigations have been reported. The investigators are going to find out if Hartmann's solution actually raises postoperative glucose and insulin level by comparing two groups of diabetic patients using either Hartmann's solution or normal saline. The investigators expect the result to broaden the choice of fluid for diabetic patients undergoing surgery and hopefully to diminish the side effects manifested by the excess use of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes patients who are included in American Society of Anesthesiologists Physical Status Classification I-III.

Exclusion Criteria:

* emergency surgery, acute or chronic kidney disease, electrolyte imbalance such as hypernatremia, hyponatremia, hyperkalemia or hypokalemia, liver dysfunction, unexpected hemodynamic instability due to excess bleeding, postoperative ventilatory care and trauma patients.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative glucose level | up to postoperative day 2
  Being the first blood sampling done a day before the surgery as the baseline, postoperative blood glucose levels checked at one hour after the surgery, and first and second postoperative days

SECONDARY OUTCOMES:
Postoperative Stress hormone level | up to postoperative day 2
  Insulin, Glucagon, Free Fatty Acid, Cortisol, Lactate, Ketone body are checked at one hour after the surgery, and first and second postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, MD, Principal Investigator — Yeungnam University College of Medicine
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

REFERENCES:
- [Background] Wolfe RR, Allsop JR, Burke JF. Glucose metabolism in man: responses to intravenous glucose infusion. Metabolism. 1979 Mar;28(3):210-20. doi: 10.1016/0026-0495(79)90066-0. PMID 763155
- [Result] Sato T, Hoshi H, Kumon T, Kitakaze Y, Watanabe R, Kobayashi T, Yoshinaga K. Managing diabetic surgical patients with glucose-free saline and insulin. Diabetes Res Clin Pract. 1988 Sep 5;5(3):191-5. doi: 10.1016/s0168-8227(88)80087-1. PMID 3065017
- See also: Glucose metabolism in man: responses to intravenous glucose infusion — http://www.ncbi.nlm.nih.gov/pubmed/763155
- See also: Managing diabetic surgical patients with glucose-free saline and insulin — http://www.ncbi.nlm.nih.gov/pubmed/3065017